CLINICAL TRIAL: NCT00032357
Title: CSP #410 - The Iron (Fe) and Atherosclerosis Study (FeAST)
Brief Title: Does the Reduction of Total Body Iron Storage (TBIS) Alter Mortality in a Population of Patients With Advanced PVD?
Acronym: FeAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 410
Record Dates: First submitted 2002-03-19; First posted 2002-03-20 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Atherosclerosis; Intermittent Claudication; Peripheral Vascular Diseases
Keywords: Ferritin reduction; Peripheral Vascular Disease (PVD); phlebotomy; Reduction of Total Body Iron Storage(TBIS); Total Body Iron Storage(TBIS)
MeSH Terms: conditions — Atherosclerosis; Intermittent Claudication; Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Other): Usual care plus Ferritin reduction to a calculated nadir of 25 ng/mL by phlebotomy
  Interventions: Procedure: Ferritin reduction to 25 ng/ml by phlebotomy
- Arm 2 (No Intervention): Usual care only; no intervention control

INTERVENTIONS:
Procedure: Ferritin reduction to 25 ng/ml by phlebotomy
  Arms: Arm 1

SUMMARY:
Veterans Affairs Cooperative Study #410, The Iron and Atherosclerosis Trial, FeAST, a 24-hospital prospective randomized single-blinded clinical trial of graded iron reduction was conducted between May 1, 1999 and April 30, 2005, and has now been completed. A total of 1,277 primarily male participants with peripheral arterial disease were entered. The primary outcome was all cause mortality and the secondary outcome combined death plus non-fatal myocardial infarction (MI) and stroke.

DETAILED DESCRIPTION:
The original JAMA abstract (2007) reported no overall effect of iron reduction intervention by phlebotomy. However, pre-planned analyses according to randomization variables at entry, including age and ferritin level, were described in the JAMA paper showing improved outcomes with iron reduction with younger age by quartile for the secondary endpoint (p for interaction =0.004) and also suggested a favorable effect in smokers (p for interaction 0.006). Age analyzed as a continuous variable using the Cox proportional hazards regression model and log relative hazard plots revealed that age interacted nonlinearly with treatment in both primary (p=0.04) and secondary (p<0.001) outcomes. The Cox model showed improved primary (HR 0.47, 95% CI 0.24-0.90, p=0.02) and secondary (HR 0.41, 95% CI 0.24-0.68, p<0.001) outcomes in youngest age quartile participants (age 43 to 61) randomized to iron reduction versus control. Thus, an interaction between age and level of body iron may have masked beneficial effects of iron reduction in the overall cohort.

Detailed analysis of the effect of age and ferritin levels published in the American Heart Journal confirmed that iron reduction significantly improved primary and secondary outcomes in youngest age quartile participants, as described above, displayed as Kaplan-Meier plots. Mean follow-up ferritin levels (MFFL) declined with increasing entry age in controls. Older age (p=0.026) and higher ferritin (p<0.001) at entry predicted poorer compliance with phlebotomy and rising MFFL in iron reduction participants. Iron reduction intervention also produced greater ferritin reduction in younger participants. Improved outcomes with lower MFFL occurred in iron reduction patients for both primary (HR 1.11, 95% CI 1.01-1.23, p=0.028) and secondary (HR 1.10, 95% CI 1.0-1.20, p=0.044) outcomes, and for the entire cohort: primary outcome (HR 1.11, 95% CI 1.01-1.23, p=0.037). Improved outcomes occurred with MFFL below versus above the median of the entire cohort means: primary outcome HR 1.48, 95% CI 1.14-1.92, p=0.003; secondary outcome HR 1.22, 95% CI 0.99-1.50, p=0.067.

Thus, lower iron burden predicted improved outcomes overall and was enhanced with iron reduction by phlebotomy. Controlling iron burden may improve survival, and prevent or delay non-fatal myocardial infarction and stroke. These findings warrant confirmation using further studies.

A possible effect of iron levels on risk of cancer as well as vascular disease was recognized at trial inception. Participants with visceral malignancy within the preceding five years were excluded from this study. However, information was collected prospectively on the occurrence of new visceral malignancy and cause-specific mortality including death due to cancer. As reported in the Journal of the National Cancer Institute, a new visceral malignancy was diagnosed during follow-up in 60 control and 38 iron reduction participants, a 37% (HR 0.63; 95% CI = 0.42 - 0.95, p = 0.026) decrease in risk with iron reduction. Reduced cancer risk with iron reduction was confirmed on time-to-event analysis (HR = 0.65; 95% CI = 0.43 - 0.97, p = 0.036). Reduced risk was observed for several common tumor types. Iron reduction participants had lower cancer - specific mortality and lower all-cause mortality in participants diagnosed with cancer (HR = 0.39; 95% CI = 0.21 - 0.72, p = 0.003 and HR = 0.49; 95% CI = 0.29 - 0.83, p = 0.009 respectively), compared to control participants. MFFL during follow-up in those participants randomized to iron reduction who developed cancer were comparable to levels in control participants (t93 = 0.8, p = 0.428). The MFFL in participants randomized to iron reduction developing cancer was 127 ng/mL, 95% CI = 71.2 - 183.0. The MFFL was significantly lower in participants not developing cancer, 76.4 ng/mL, 95% CI = 71.4 - 81.4, p = 0.017). Participants randomized to iron reduction developing cancer appeared to be relatively non-compliant with intervention.

Analysis of data from the FeAST study continues to delineate interactions between iron status and smoking, lipid levels and statin use, diabetes and race. It has been shown that ferritin levels ranging from about 70 to 79 ng/mL are associated with lower mortality and levels of inflammatory markers. Statin use, while not a randomization variable, has been monitored and shown to relate to lower ferritin levels.

ELIGIBILITY:
Inclusion Criteria:

1. Males over the age of 21 years and post menopausal (either natural or surgical) females with a diagnosis of intermittent claudication who are not scheduled for major surgery and who can give informed consent will be entered.
2. Hematocrit of 30% or greater for females and 35% or greater for males, normal liver function, serum creatinine less than 4 mg/dl. Patients with mild anemia and mild creatinine elevation will be entered (provided the anemia is not due to Fe deficiency found on screening laboratory tests) because such findings are commonly present chronically in PVD.
3. Absence of a disturbance in Fe balance (e.g. hemosiderosis from any cause, hemochromatosis, atransferrinemia, PNH, Fe deficiency)
4. Absence for at least six months of a disease that has caused bleeding (e.g. peptic ulcer, inflammatory bowel disease, hemorrhagic diathesis )
5. Absence of associated neoplasm other than epithelial ( non-melanoma) tumors of skin or other co-morbid condition that is expected to be fatal within one year.
6. Absence of an associated obvious inflammatory disorder (e.g. infection, connective tis-sue disease) capable of elevating ferritin levels acutely.
7. Patients will not be excluded on the basis of either the existence or severity of either coronary- or cerebrovascular disease, medication use including non-steroidal anti-inflammatory drugs and anticoagulants, coronary angiographic findings, previous history of or possible future need for angioplasty or coronary bypass surgery, or elevated blood pressure.
8. Patients must agree to not take any Fe supplements or vitamins while on study.

Exclusion Criteria:

1. Patients must have at least one lower extremity and must not be on another experimental therapy protocol for atherosclerotic vascular disease.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1277 (Actual)
Dates: Start 1999-05; Primary Completion 2005-04 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Mortality | The minimum follow-up was 3.5 years and maximum follow-up was 6 years
  The primary objective of this study is to evaluate the effectiveness of a reduction of Total Body Iron Stores (TBIS) in decreasing the rate of all cause mortality in patients with peripheral vascular disease (PVD).

CONTACTS AND LOCATIONS:
Overall Officials: Zacharski R. Leo, Study Chair — VA Medical & Regional Office Center, White River
Locations (24):
- United States (23):
  - VA Medical Center, Birmingham, Birmingham, Alabama
  - Central Arkansas VHS Eugene J. Towbin Healthcare Ctr, Little Rock, No. Little Rock, Arkansas
  - VA Medical Center, Long Beach, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - VA Connecticut Health Care System (West Haven), West Haven, Connecticut
  - North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - James A. Haley Veterans Hospital, Tampa, Tampa, Florida
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - VA Medical Center, Lexington, Lexington, Kentucky
  - VA Medical Center, Louisville, Louisville, Kentucky
  - VA Medical Center, Jamaica Plain Campus, Boston, Massachusetts
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - VA Stratton Medical Center, Albany, Albany, New York
  - New York Harbor HCS, New York, New York
  - VA Medical Center, Durham, Durham, North Carolina
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania
  - VA Medical Center, Providence, Providence, Rhode Island
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, Salt Lake City, Utah
  - VA Medical & Regional Office Center, White River, White River Junction, Vermont
  - Wlliam S. Middleton Memorial Veterans Hospital, Madison, Madison, Wisconsin
  - Zablocki VA Medical Center, Milwaukee, Milwaukee, Wisconsin
- VA Medical Center, San Juan, San Juan, Puerto Rico

REFERENCES:
- [Result] DePalma RG, Hayes VW, Cafferata HT, Mohammadpour HA, Chow BK, Zacharski LR, Hall MR. Cytokine signatures in atherosclerotic claudicants. J Surg Res. 2003 May 15;111(2):215-21. doi: 10.1016/s0022-4804(03)00075-1. PMID 12850465
- [Result] DePalma RG, Hayes VW, May PE, Cafferata HT, Mohammadpour HA, Brigg LA, Chow BK, Shamayeva G, Zacharski LR. Statins and biomarkers in claudicants with peripheral arterial disease: cross-sectional study. Vascular. 2006 Jul-Aug;14(4):193-200. doi: 10.2310/6670.2006.00039. PMID 17026909
- [Result] Zacharski LR, Chow BK, Howes PS, Shamayeva G, Baron JA, Dalman RL, Malenka DJ, Ozaki CK, Lavori PW. Reduction of iron stores and cardiovascular outcomes in patients with peripheral arterial disease: a randomized controlled trial. JAMA. 2007 Feb 14;297(6):603-10. doi: 10.1001/jama.297.6.603. PMID 17299195
- [Result] DePalma RG, Hayes VW, Zacharski LR. Bloodletting: past and present. J Am Coll Surg. 2007 Jul;205(1):132-44. doi: 10.1016/j.jamcollsurg.2007.01.071. Epub 2007 May 17. No abstract available. PMID 17617342
- [Result] Depalma RG, Hayes VW, Chow BK, Shamayeva G, May PE, Zacharski LR. Ferritin levels, inflammatory biomarkers, and mortality in peripheral arterial disease: a substudy of the Iron (Fe) and Atherosclerosis Study (FeAST) Trial. J Vasc Surg. 2010 Jun;51(6):1498-503. doi: 10.1016/j.jvs.2009.12.068. Epub 2010 Mar 20. PMID 20304584
- [Result] Depalma RG, Zacharski LR. Iron reduction benefits: positive results from a "negative" prospective randomized controlled trial. Vasc Endovascular Surg. 2012 Oct;46(7):596-7. doi: 10.1177/1538574412456304. Epub 2012 Aug 17. No abstract available. PMID 22903331
- [Result] Zacharski LR, Shamayeva G, Chow BK. Effect of controlled reduction of body iron stores on clinical outcomes in peripheral arterial disease. Am Heart J. 2011 Nov;162(5):949-957.e1. doi: 10.1016/j.ahj.2011.08.013. PMID 22093213
- [Result] Zacharski LR, Chow BK, Howes PS, Shamayeva G, Baron JA, Dalman RL, Malenka DJ, Ozaki CK, Lavori PW. Decreased cancer risk after iron reduction in patients with peripheral arterial disease: results from a randomized trial. J Natl Cancer Inst. 2008 Jul 16;100(14):996-1002. doi: 10.1093/jnci/djn209. Epub 2008 Jul 8. PMID 18612130
- [Result] Zacharski LR, Chow BK, Howes PS, Lavori PW, Shamayeva G. Implementation of an iron reduction protocol in patients with peripheral vascular disease: VA cooperative study no. 410: the Iron (Fe) and Atherosclerosis Study (FeAST). Am Heart J. 2004 Sep;148(3):386-92. doi: 10.1016/j.ahj.2004.03.027. PMID 15389223
- [Result] Zacharski LR, Chow B, Lavori PW, Howes PS, Bell MR, DiTommaso MA, Carnegie NM, Bech F, Amidi M, Muluk S. The iron (Fe) and atherosclerosis study (FeAST): a pilot study of reduction of body iron stores in atherosclerotic peripheral vascular disease. Am Heart J. 2000 Feb;139(2 Pt 1):337-45. doi: 10.1067/mhj.2000.102909. PMID 10650308
- [Derived] DePalma RG, Zacharski LR, Chow BK, Shamayeva G, Hayes VW. Reduction of iron stores and clinical outcomes in peripheral arterial disease: outcome comparisons in smokers and non-smokers. Vascular. 2013 Aug;21(4):233-41. doi: 10.1177/1708538113478776. PMID 23518844